CLINICAL TRIAL: NCT02624908
Title: Canagliflozin-Mealtime Insulin Rescue
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation for Atlanta Veterans Education and Research, Inc. (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28431754DIA4008
Record Dates: First submitted 2015-12-03; First posted 2015-12-09 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- canagliflozin (Active Comparator): Subjects randomized to this arm will start with 100 mg tablet and increase to 300 mg tablet at Visit 4 if well tolerated.
  Interventions: Drug: canagliflozin
- placebo (Placebo Comparator): Subjects randomized to this arm will start with 100 mg tablet and increase to 300 mg tablet at Visit 4 if well tolerated.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: canagliflozin — Subjects randomized to active drug will receive canagliflozin 100 mg . If study drug well tolerated, dose will be increased to 300 mg canagliflozin at Visit 4.
  Other Names: Invokana
  Arms: canagliflozin
Drug: placebo — Subjects randomized to placebo will receive 100 mg placebo pill . If study drug well tolerated, dose will be increased to 300 mg placebo pill at Visit 4.
  Other Names: inactive substance
  Arms: placebo

SUMMARY:
24-week, randomized, double blind, placebo-controlled trial to evaluate safety and efficacy of canagliflozin as compared with placebo in reducing the need for mealtime insulin in subjects with type 2 diabetes currently using a basal-bolus insulin regimen.

DETAILED DESCRIPTION:
The Canagliflozin Mealtime Insulin Rescue study will enroll up to 40 subjects at the Atlanta VA Medical Center. Subjects will be screened and enter a 2-week run-in period during which they will switch to or continue on a diabetes treatment regimen of basal insulin before supper and aspart insulin before meals. Run-in will be useful in evaluating compliance to treatment and self-monitoring. After run-in, subjects will collect one week of baseline glycemic data with regular pre-meal and fasting glycemic levels using both finger stick testing and continuous glucose monitoring.

Subjects will be randomized at Visit 3 to 100 mg of canagliflozin or placebo. If well tolerated, this dose will be increased to 300 mg of canagliflozin or placebo at Visit 4.

Diabetes management will be assured through regular contact with the study team (weekly calls and clinic visits at Weeks 4, 8, 16 and 24). Management will be facilitated by diabetes management software. Self-monitoring and continuous glucose monitoring will be repeated at the end of study participation.

ELIGIBILITY:
Inclusion Criteria:

* use of basal-bolus insulin
* onset of diabetes after age 30
* BMI less than 35
* eGFR at least 60 ml/mn
* Hb A1c 7.0-10.0%
* willingness to perform home glucose monitoring
* willingness to transmit glucose and medication information weekly

Exclusion Criteria:

* Type 1 diabetes
* Known peripheral artery disease
* Liver enzymes equal or more than 1.5 times the upper limit of normal
* Chronic heart failure NYHA class III or IV
* Current haemodialysis or peritoneal dialysis
* End stage liver disease, defined as acute or chronic liver disease and recent history of one of the following: ascites, encephalopathy, variceal bleeding, bilirubin equal or greater than 2.0 mg/dL, albumin equal or less than 3.5 g/ dL, prothrombin time greater or equal to 4 seconds, INR greater than or equal to 1.7 or prior liver transplant
* Known or suspected hypersensitivity to trial products or related products
* Female of child-bearing potential who is pregnant, breast-feeding or intends to become pregnant or is not using adequate contraceptive methods as required by law or local practice.
* Expected simultaneous participation in any other clinical trial of an investigational medicinal product.
* Receipt of any investigational medicinal product within 30 days before randomization
* Current or past (within the last 5 years) malignant neoplasms (except basal cell and squamous cell skin carcinoma)
* Any condition that in the investigator's opinion would make the subject unable to adhere to the trial visit schedule and procedures
* Known history of non-compliance to treatment.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients who discontinue all pre-meal medications for at least one meal per day | 24 weeks
Number of patients who replace mealtime insulin with an oral agent for at least one meal per day | 24 weeks
  anti-hyperglycemic pill instead of insulin for at least one meal per day
Number of patients with a continuing need for insulin 4 times per day | 24 weeks
  no change from the original basal -bolus regimen
Frequency and severity of hypoglycemia | 24 weeks
  Hypoglycemic episodes will be evaluated using a hypoglycemia questionnaire
Self monitoring and continuous monitoring blood glucose levels | 24 weeks
  glycemic control and glycemic variability

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence S Phillips, MD, Principal Investigator — Atlanta VA Medical Center
Locations (1):
- Atlanta VA Medical Center, Decatur, Georgia, United States

REFERENCES:
- [Background] ORIGIN Trial Investigators; Gerstein HC, Bosch J, Dagenais GR, Diaz R, Jung H, Maggioni AP, Pogue J, Probstfield J, Ramachandran A, Riddle MC, Ryden LE, Yusuf S. Basal insulin and cardiovascular and other outcomes in dysglycemia. N Engl J Med. 2012 Jul 26;367(4):319-28. doi: 10.1056/NEJMoa1203858. Epub 2012 Jun 11. PMID 22686416
- [Background] Bretzel RG, Nuber U, Landgraf W, Owens DR, Bradley C, Linn T. Once-daily basal insulin glargine versus thrice-daily prandial insulin lispro in people with type 2 diabetes on oral hypoglycaemic agents (APOLLO): an open randomised controlled trial. Lancet. 2008 Mar 29;371(9618):1073-84. doi: 10.1016/S0140-6736(08)60485-7. PMID 18374840
- [Background] Schernthaner G, Gross JL, Rosenstock J, Guarisco M, Fu M, Yee J, Kawaguchi M, Canovatchel W, Meininger G. Canagliflozin compared with sitagliptin for patients with type 2 diabetes who do not have adequate glycemic control with metformin plus sulfonylurea: a 52-week randomized trial. Diabetes Care. 2013 Sep;36(9):2508-15. doi: 10.2337/dc12-2491. Epub 2013 Apr 5. PMID 23564919
- [Background] Polidori D, Sha S, Mudaliar S, Ciaraldi TP, Ghosh A, Vaccaro N, Farrell K, Rothenberg P, Henry RR. Canagliflozin lowers postprandial glucose and insulin by delaying intestinal glucose absorption in addition to increasing urinary glucose excretion: results of a randomized, placebo-controlled study. Diabetes Care. 2013 Aug;36(8):2154-61. doi: 10.2337/dc12-2391. Epub 2013 Feb 14. PMID 23412078
- [Background] Budnitz DS, Lovegrove MC, Shehab N, Richards CL. Emergency hospitalizations for adverse drug events in older Americans. N Engl J Med. 2011 Nov 24;365(21):2002-12. doi: 10.1056/NEJMsa1103053. PMID 22111719
- [Background] Home PD, Fritsche A, Schinzel S, Massi-Benedetti M. Meta-analysis of individual patient data to assess the risk of hypoglycaemia in people with type 2 diabetes using NPH insulin or insulin glargine. Diabetes Obes Metab. 2010 Sep;12(9):772-9. doi: 10.1111/j.1463-1326.2010.01232.x. PMID 20649629
- [Background] Johnston SS, Conner C, Aagren M, Smith DM, Bouchard J, Brett J. Evidence linking hypoglycemic events to an increased risk of acute cardiovascular events in patients with type 2 diabetes. Diabetes Care. 2011 May;34(5):1164-70. doi: 10.2337/dc10-1915. Epub 2011 Mar 18. PMID 21421802
- [Background] NICE-SUGAR Study Investigators; Finfer S, Liu B, Chittock DR, Norton R, Myburgh JA, McArthur C, Mitchell I, Foster D, Dhingra V, Henderson WR, Ronco JJ, Bellomo R, Cook D, McDonald E, Dodek P, Hebert PC, Heyland DK, Robinson BG. Hypoglycemia and risk of death in critically ill patients. N Engl J Med. 2012 Sep 20;367(12):1108-18. doi: 10.1056/NEJMoa1204942. PMID 22992074
- [Background] McCoy RG, Van Houten HK, Ziegenfuss JY, Shah ND, Wermers RA, Smith SA. Increased mortality of patients with diabetes reporting severe hypoglycemia. Diabetes Care. 2012 Sep;35(9):1897-901. doi: 10.2337/dc11-2054. Epub 2012 Jun 14. PMID 22699297
- [Background] Ceriello A, Esposito K, Piconi L, Ihnat MA, Thorpe JE, Testa R, Boemi M, Giugliano D. Oscillating glucose is more deleterious to endothelial function and oxidative stress than mean glucose in normal and type 2 diabetic patients. Diabetes. 2008 May;57(5):1349-54. doi: 10.2337/db08-0063. Epub 2008 Feb 25. PMID 18299315
- [Background] Brownlee M, Hirsch IB. Glycemic variability: a hemoglobin A1c-independent risk factor for diabetic complications. JAMA. 2006 Apr 12;295(14):1707-8. doi: 10.1001/jama.295.14.1707. No abstract available. PMID 16609094